CLINICAL TRIAL: NCT01524575
Title: Phase II Study of Gemcitabine and Oxaliplatin in the Management of Metastatic Pancreatic Cancers With Low Expression of ERCC1 (Excision Repair Cross-complementation Group 1)
Brief Title: Gemcitabine and Oxaliplatin in the Management of Metastatic Pancreatic Cancers With Low Expression of ERCC1
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: the trial was never opened and then withdrawn permanently
Sponsor: University of Hawaii (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRCH0904
Record Dates: First submitted 2012-01-26; First posted 2012-02-02 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Metastatic Pancreatic Cancer; ERCC1
Keywords: pancreatic cancer; ERCC1; oxaliplatin; gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ERCC1 high expression (No Intervention): Patients with ERCC1 high expression tumors will be treated at discretion of investigator
- ERCC1 low expression (Experimental): Patients with ERCC1 low expression will be treated with gemcitabine and oxaliplatin
  Interventions: Drug: gemcitabine and oxaliplatin

INTERVENTIONS:
Drug: gemcitabine and oxaliplatin — Excision repair cross-complementation group 1 (ERCC1) protein and mRNA expression predicts response to oxaliplatin - patients whose cancers make small amounts of ERCC1 are much more likely to respond to cisplatin than those whose tumors produce large amounts.
  Other Names: gemcitabine 1000mg/m2 IV q2week and oxaliplatin 85mg/m2 IV q2week
  Arms: ERCC1 low expression

SUMMARY:
The goal of this clinical trial is to improve and personalize pancreatic cancer care to deliver the most effective therapy while avoiding unnecessary exposure to potential side effects. Excision repair cross-complementation group 1 (ERCC1) protein and mRNA expression predicts response to oxaliplatin - patients whose cancers make small amounts of ERCC1 are much more likely to respond to cisplatin than those whose tumors produce large amounts. The hypothesis is that the combination of gemcitabine and oxaliplatin is a uniquely effective regimen for patients with metastatic pancreatic cancer whose tumors have a low expression of ERCC1.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic pancreatic adenocarcinoma
* Patients must not have had prior chemotherapy or biologic therapy for metastatic pancreatic cancer
* Prior adjuvant chemotherapy for completely resected disease or chemoradiotherapy for locally advanced disease is allowed but must have been administered > 6 months prior to registration
* ECOG Performance Status of 0, 1, or 2
* Adequate hematologic, hepatic and renal function

Exclusion Criteria:

* Pregnant or nursing women
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or any other cancer from which the patient has been disease-free for 5 years
* Patients must not have known brain metastases
* Any other condition that in the opinion of the Investigator may render the patient at excessive risk for treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01 (Estimated); Primary Completion 2013-07 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
6 month overall survival | 6 months

SECONDARY OUTCOMES:
Overall survival | Assessments every 2 months until 2 years or death
Progression free survival | Assessments every 2 months with CT scan until progression by RECIST criteria up to maximum of 2 years
Best confirmed response | Assessments every 2 months with CT scan until progression by RECIST criteria up to maximum of 2 years
Duration of overall response | Assessments every 2 months with CT scan until progression by RECIST criteria up to maximum of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jared D Acoba, MD, Principal Investigator — University of Hawaii Cancer Research Center
Locations (1):
- University of Hawaii, Honolulu, Hawaii, United States